CLINICAL TRIAL: NCT05955573
Title: What Affects the Severity of Knee Osteoarthritis? Aging or Associated Metabolic Syndrome
Brief Title: Knee Osteoarthritis, Aging and Metabolic Syndrome
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amany Mohamed Abdelrahman, Physical Medicine, Rheumatology and Rehabilitation Department, Sohag University
Other Study IDs: Soh-Med-23-07-17MS
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; Aging; Metabolic Syndrome
MeSH Terms: conditions — Osteoarthritis, Knee; Metabolic Syndrome | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- knee osteoarthritis: Knee osteoarthritis
  Interventions: Diagnostic Test: xray

INTERVENTIONS:
Diagnostic Test: xray — radiological description

SUMMARY:
Osteoarthritis (OA) is the most prevalent form of arthritis. Its pathogenesis remains poorly understood. Though historically regarded as a disease of mechanical degeneration, it is now appreciated that inflammation plays an important role in OA pathogenesis

DETAILED DESCRIPTION:
1. Place of the study: Sohag university hospital.
2. Type of study: Cross-Sectional Observational study
3. Study period: Six months to one year The study will include Patients who met the American College of Rheumatology (ACR) clinical criteria for knee OA .

The following details will be obtained:

* Demographic data : Age ,Sex ,Marital status ,Occupation ,Residence ,Education level

  ,Anthropometrical measures which included waist circumference (WC) and blood pressure (BP) will be obtained,History of chronic diseases (eg; Diabetes mellites, Hypertension)
* Clinical information: Symptom and its Duration. Plain radiographs of at least one knee [anteroposterior (A/P), lateral} will be taken.
* Laboratory findings included fasting blood sugar, serum levels of triglycerides, High-density lipoprotein cholesterol and total cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met the American College of Rheumatology (ACR) clinical criteria for knee OA and had symptomatic OA of at least 1 knee (index knee), with a Kellgren / Lawrence (K/L) score ≥ 1 in that knee

Exclusion Criteria:

* Any patient with a history of trauma to the knee

  * Any other form of arthritis (e.g., rheumatoid arthritis, seronegative spondyloarthropathies, gout, pyrophosphate disease, or other crystal arthropathy)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: knee osteoartgritis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
severity of knee osteoarthritis | 8/2023-8/2024
  Kellgren and Lawrence (K/L) grading system of Knee osteoarthritis. It assigned a grade from 0 to 4, which they correlated to increasing severity of OA, with Grade 0 signifying no presence of OA and Grade 4 signifying severe OA .

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Shaker Elgendy, MD, Study Chair — Sohag University; Hanan Sayed Abo-zaid, MD, Study Director — Sohag University
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Englund, M. (202+3). Osteoarthritis, part of life or a curable disease? A bird's-eye view. In Journal of Internal Medicine. John Wiley and Sons Inc. https://doi.org/10.1111/joim.13634 Grundy, S. M., Cleeman, J. I., Daniels, S. R., Donato, K. A., Eckel, R. H., Franklin, B. A., Gordon, D. J., Krauss, R. M., Savage, P. J., Smith, S. C., Spertus, J. A., & Costa, F. (2005). Diagnosis and management of the metabolic syndrome: An American Heart Association/National Heart, Lung, and Blood Institute scientific statement. In Circulation (Vol. 112, Issue 17, pp. 2735-2752). https://doi.org/10.1161/CIRCULATIONAHA.105.169404 KELLGREN, J. H., & LAWRENCE, J. S. (1957). Radiological assessment of osteo-arthrosis. Annals of the Rheumatic Diseases, 16(4), 494-502. https://doi.org/10
- [Background] Krasnokutsky S, Oshinsky C, Attur M, Ma S, Zhou H, Zheng F, Chen M, Patel J, Samuels J, Pike VC, Regatte R, Bencardino J, Rybak L, Abramson S, Pillinger MH. Serum Urate Levels Predict Joint Space Narrowing in Non-Gout Patients With Medial Knee Osteoarthritis. Arthritis Rheumatol. 2017 Jun;69(6):1213-1220. doi: 10.1002/art.40069. Epub 2017 Apr 28. PMID 28217895
- See also: Related Info — https://doi.org/10.1038/s41598-023-30727-4